CLINICAL TRIAL: NCT01013142
Title: A Phase I Randomized, Double-blind, Placebo-controlled Dose Escalation Study to Evaluate the Safety and Efficacy of MN-221 When Administered Intravenously to Subjects With Stable Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Evaluate the Safety of MN-221 in Subjects With Stable Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MN-221-CL-010
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — bedoradrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MN-221 (Experimental)
  Interventions: Drug: MN-221 (Dose Group 1); Drug: MN-221 (Dose Group 2); Drug: MN-221 (Dose Group 3)
- MN-221 Placebo (Placebo Comparator)
  Interventions: Drug: MN-221 (Dose Group 1); Drug: MN-221 (Dose Group 2); Drug: MN-221 (Dose Group 3)

INTERVENTIONS:
Drug: MN-221 (Dose Group 1) — i.v. infusion of MN-221 (300 mcg) or placebo over 1 hour
Drug: MN-221 (Dose Group 2) — i.v. infusion of MN-221 (600 mcg) or placebo over 1 hour
Drug: MN-221 (Dose Group 3) — i.v. infusion of MN-221 (1,200 mcg) or placebo over 1 hour

SUMMARY:
The objective of this clinical study is to determine the safety of intravenous MN-221 compared to placebo when administered in subjects diagnosed with stable moderate to severe COPD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center dose escalation study in subjects diagnosed with stable moderate to severe COPD. The study will be conducted in approximately 6 Clinical Research Units (CRUs).

Subjects with a diagnosis of stable moderate to severe COPD will be screened and must demonstrate an improvement in FEV1 after bronchodilator treatment of at least 12% at Screen Visit 1. The subject's degree of dyspnea will be captured on the British Medical Research Council (MRC) questionnaire, and severity will be determined by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) spirometric criteria. Subjects meeting entry criteria at Screen Visit 1 will be asked to return to the CRU for Screen Visit 2 within 14 days of Visit 1. Subjects confirming entry criteria including degree of COPD severity by spirometry at Screen Visit 2 will be randomized to receive either MN-221 or placebo. Serial spirometry will be performed over the 8 hour treatment period after initiation of study drug administration. Subjects will be discharged from the CRU after completing the Hour 8 study procedures and asked to return approximately 24 hours after initiation of study drug for follow up safety assessments including spirometry. A study diary will be provided to each subject upon discharge from the CRU to complete as instructed and return it to the site at the 24 hour Follow-up Visit.

There will be three dose levels and each will include approximately 16 subjects randomized to receive either MN-221 or placebo in 3:1 ratio (12 subjects receive MN-221:4 subjects receive placebo). A risk/benefit evaluation will be performed by the study's Safety Review Committee at completion of each dose level prior to escalating to the next dose level.

Safety and efficacy will be monitored throughout the treatment period. Blood samples for PK parameters and metabolite identification will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 40-65 years of age, inclusive;
2. History of physician-diagnosed COPD treated for ≥ 3 months ;
3. FEV1 ≥ 30% < 80% and FEV1/FVC ratio < 0.7 at screening;
4. An increase in FEV1 of at least 12%, over the pre-albuterol FEV1 within 30 minutes after inhalation of albuterol;
5. Negative urine pregnancy test for all females unless the subject is post-menopausal (≥ 24 months of spontaneous amenorrhea) or surgically sterile (hysterectomy, bilateral ovariectomy or bilateral tubal ligation);
6. Negative urine drug screen for cocaine, PCP, methamphetamine;
7. ECG with no evidence of ischemic heart disease or dysrhythmias and otherwise normal or with findings considered not clinically significant at screening;
8. QTcB and QTcF < 450 msec;
9. No clinical evidence of active ischemic heart disease as determined by the Investigator; and
10. Legally effective written informed consent obtained prior to starting any study procedures.

Exclusion Criteria:

1. Beta agonist and/or anticholinergic via inhaler or intravenously ≤ 6 hours of screening;
2. Sustained release methylxanthine (e.g. Theophylline) or long acting beta agonists ≤ 24 hours prior to screening;
3. A diagnosis of clinically significant myocardial or valvular disease; including cardiomyopathy, congestive heart failure, or pulmonary edema;
4. Acute exacerbation of COPD requiring emergency treatment ≤ 30 days of screening or hospitalization ≤ 90 days of screening;
5. Antibiotic therapy for respiratory infection ≤ 30 days of screening;
6. Presence of active respiratory disease such as pneumonia, or acute bronchitis;
7. History or presence of tachyarrhythmias, with the exception of sinus tachycardia;
8. Hypokalemia defined as a potassium level ≤ 3.0 mmol/L at screening;
9. Significant renal, hepatic, endocrine, metabolic, neurologic or other systemic disease;
10. Uncontrolled hypertension defined as a blood pressure ≥ 170/100 mm Hg at screening;
11. Pregnant or lactating females;
12. Participation in another clinical study with an investigational drug within 30 days of screening;
13. A known allergy to excipients of the MN-221 drug product;
14. A known allergy to other beta agonists;
15. Previous exposure to MN-221; or
16. Use of beta blockers, MAO inhibitors, or tricyclic antidepressants ≤ 2 weeks prior to screening.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Adverse events, cardiac and ECG parameters, vital signs, physical exam and clinical laboratory assessments. | Hour 0 (treatment) through Hour 24 (follow-up)

SECONDARY OUTCOMES:
Pharmacokinetic parameters of MN-221. | Pre-dose to Hour 24 post-dose
Forced expiratory volume in one second (FEV1). | Pre-dose to Hour 24 post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Alan W Dunton, MD, Study Director — MediciNova
Locations (7):
- United States (7):
  - Dedicated Phase I, Phoenix, Arizona
  - California Research Medical Group, INC, Fullerton, California
  - Vita Research Solutions & Medical Center, Inc., Tamarac, Florida
  - Florida Pulmonary Research Institue, LLC, Winter Park, Florida
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Gulf Coast Research, LLC, Lafayette, Louisiana
  - SNBL CLinical Pharmacology Center, Baltimore, Maryland